CLINICAL TRIAL: NCT03120988
Title: Assessing Catabolic Marker Levels in the Knee Synovial Fluid Microenvironment After Lavage With Platelet Poor Plasma (PPP)
Brief Title: Catabolic Marker Levels After Platelet Poor Plasma (PPP) Lavage
Acronym: PPP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSI2015-LAB03
Record Dates: First submitted 2016-12-19; First posted 2017-04-19 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee OA; lavage; Platelet Poor Plasma (PPP)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: Lavage with platelet poor plasma
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lavage with Platelet Poor Plasma (PPP) (Experimental): Lavage using 50 cc of PPP in the knee joint. Using visual guidance, the PPP lavage will be conducted, introducing a solution of platelet poor plasma into the knee joint with subsequent removal of the fluid, in effect "washing out" the joint space.
  Interventions: Biological: Lavage with Platelet Poor Plasma (PPP)

INTERVENTIONS:
Biological: Lavage with Platelet Poor Plasma (PPP) — Lavage of 50cc PPP

SUMMARY:
The purpose of this study is to understand how the components of osteoarthritic knee joint fluid (synovial fluid) change after lavage treatment with platelet poor plasma. Additionally, the study participants will complete outcome questionnaire surveys before and after the treatment in conjunction with when synovial fluid is removed from the knee (2, 4, and 6 weeks after lavage). This data will help determine if the treatment of an osteoarthritic knee joint with platelet poor plasma lavage is a suitable stand-alone therapy or to improve outcome by preparing a patient's knee for further regenerative therapies.

DETAILED DESCRIPTION:
The objective of this study is to quantify the levels of catabolic markers in osteoarthritic (OA) knee synovial fluid microenvironment (ME) before lavage treatment with platelet poor plasma (PPP) and to determine whether the anti-catabolic capabilities of the PPP are sustainable or if the diseased synovial fluid returns to pre-lavage catabolic marker levels within the 6 week period of the study.

This data will be used to determine if treatment of a diseased (OA) knee with PPP lavage would be a suitable therapy for knee OA patients either as a stand-alone treatment or to improve outcome by preparing a patient's knee microenvironment for further treatment with cellular therapies. Incidence of post-operative complications, adverse events, re-injections, and surgical intervention; change in pain score will be considered while determining these direct and indirect associations upon completion of the PPP lavage treatment. Correlation of subject reported clinical outcomes for the PPP lavage treatment will be evaluated to determine whether the treatment provides beneficial clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntary signature of the institutional review board approved Informed Consent
* 2) Male or female ages 35-85
* 3) Pain, swelling, and/or functional disability in the affected knee consistent with osteoarthritis in the knee joint
* 4) Physical examination consistent with osteoarthritis as observed on imaging
* 5) Unilateral or bilateral Kellgren-Lawrence grade 3 or greater knee osteoarthritis (moderate to severe OA) and/or diagnostic MRI imaging of the affected knee showing osteoarthritis (i.e. chondral loss, fissuring, defect, bone marrow lesion, meniscus tear, synovial thickening, etc…)
* 6) Mild effusion upon ultrasound evaluation.
* 7) Is independent, ambulatory, and can comply with all postoperative evaluations and visits

Exclusion Criteria:

* 1) Knee injections of any type within 3 months prior to the study.
* 2) Knee surgery within 6 months prior to the study.
* 3) Inflammatory or auto-immune based joint diseases or other lower extremity pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
* 4) Quinolone or Statin induced myopathy/tendinopathy
* 5) Severe neurogenic inflammation of the cutaneous nerves about the knee or thigh
* 6) Contraindications for MRI
* 7) Condition represents a worker's compensation case
* 8) Currently involved in a health-related litigation procedure
* 9) Is pregnant
* 10) Bleeding disorders
* 11) Currently taking anticoagulant or immunosuppressive medication
* 12)Allergy or intolerance to study medication
* 13)Use of chronic opioid
* 14)Documented history of drug abuse within six months of treatment
* 15)Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Mean temporal biomarkers (pg/ml) | 4 weeks post treatment

SECONDARY OUTCOMES:
Mean Pain Scales | 2, 4 and 6 weeks post treatment
Mean International Knee Documentation Committee Subjective Knee Evaluation | 2, 4 and 6 weeks post treatment
Complications and adverse events | 2, 4 and 6 weeks post treatment
Mean temporal biomarkers (pg/ml) | 2 and 6 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Regenexx and Centeno-Schultz Clinic
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of doctor-diagnosed arthritis and arthritis-attributable activity limitation--United States, 2010-2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 8;62(44):869-73. PMID 24196662
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Waimann CA, Fernandez-Mazarambroz RJ, Cantor SB, Lopez-Olivo MA, Zhang H, Landon GC, Siff SJ, Suarez-Almazor ME. Cost-effectiveness of total knee replacement: a prospective cohort study. Arthritis Care Res (Hoboken). 2014 Apr;66(4):592-9. doi: 10.1002/acr.22186. PMID 24124052
- [Background] Katz JN, Brophy RH, Chaisson CE, de Chaves L, Cole BJ, Dahm DL, Donnell-Fink LA, Guermazi A, Haas AK, Jones MH, Levy BA, Mandl LA, Martin SD, Marx RG, Miniaci A, Matava MJ, Palmisano J, Reinke EK, Richardson BE, Rome BN, Safran-Norton CE, Skoniecki DJ, Solomon DH, Smith MV, Spindler KP, Stuart MJ, Wright J, Wright RW, Losina E. Surgery versus physical therapy for a meniscal tear and osteoarthritis. N Engl J Med. 2013 May 2;368(18):1675-84. doi: 10.1056/NEJMoa1301408. Epub 2013 Mar 18. PMID 23506518
- [Background] Getgood A, Collins B, Slynarski K, Kurowska E, Parker D, Engebretsen L, MacDonald PB, Litchfield R. Short-term safety and efficacy of a novel high tibial osteotomy system: a case controlled study. Knee Surg Sports Traumatol Arthrosc. 2013 Jan;21(1):260-9. doi: 10.1007/s00167-011-1709-4. Epub 2011 Oct 18. PMID 22005964
- [Background] Goldring MB, Otero M. Inflammation in osteoarthritis. Curr Opin Rheumatol. 2011 Sep;23(5):471-8. doi: 10.1097/BOR.0b013e328349c2b1. PMID 21788902
- [Background] Wang S, Wei X, Zhou J, Zhang J, Li K, Chen Q, Terek R, Fleming BC, Goldring MB, Ehrlich MG, Zhang G, Wei L. Identification of alpha2-macroglobulin as a master inhibitor of cartilage-degrading factors that attenuates the progression of posttraumatic osteoarthritis. Arthritis Rheumatol. 2014 Jul;66(7):1843-53. doi: 10.1002/art.38576. PMID 24578232
- [Background] Rehman AA, Ahsan H, Khan FH. alpha-2-Macroglobulin: a physiological guardian. J Cell Physiol. 2013 Aug;228(8):1665-75. doi: 10.1002/jcp.24266. PMID 23086799
- [Background] Irrgang JJ, Anderson AF, Boland AL, Harner CD, Neyret P, Richmond JC, Shelbourne KD; International Knee Documentation Committee. Responsiveness of the International Knee Documentation Committee Subjective Knee Form. Am J Sports Med. 2006 Oct;34(10):1567-73. doi: 10.1177/0363546506288855. Epub 2006 Jul 26. PMID 16870824